CLINICAL TRIAL: NCT00605709
Title: Dose-Ranging Safety and Efficacy Study of Topical Creams Containing API 31510 for the Treatment of in Situ Cutaneous Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Armanda Waddington/Administrative Manager, Cytotech Labs, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTL0208
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Active Cream 3% ; AM & PM
  Interventions: Drug: API 31510 Topical Cream
- 2 (Active Comparator): Placebo Cream AM; 3% Active Cream PM
  Interventions: Drug: API 31510 Topical Cream
- 3 (Active Comparator): Placebo Cream AM; 1.5% Active Cream PM
  Interventions: Drug: API 31510 Topical Cream
- 4 (Placebo Comparator): Placebo Cream AM & PM
  Interventions: Drug: API 31510 Topical Cream

INTERVENTIONS:
Drug: API 31510 Topical Cream — Topical treatments to lesion twice daily of randomized treatments.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of pharmaceutical compound 31510 in a topical cream when applied to in situ cutaneous squamous cell carcinoma and to obtain preliminary efficacy data for the treatment of in situ cutaneous squamous cell carcinoma by Compound 31510 topical cream.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ≥ 18 years of age
* Primary, histologically confirmed SCCIS with a minimum area of 0.5 cm2 and with a maximum diameter of 2.0 cm target SCCIS lesion suitable for excision
* Histological diagnosis made no more than 4 weeks prior to the screening visit
* Histological biopsy removed 25% or less of the target lesion
* No other dermatological disease in the SCCIS target site or surrounding area
* Willing to refrain from using non-approved lotions or creams on the target site and surrounding area during the treatment period. Willing to refrain from washing the treated area for at least 8 hours following the application of study medication
* Willing to refrain from exposure to direct sunlight or ultraviolet light and to avoid the use of tanning parlors for the duration of the study
* Laboratory values for the tests listed in the Study Schedule on page 2 within the reference ranges as defined by the central laboratory, or "out of range" test results that are clinically acceptable to the investigator.
* Ability to follow study instructions and likely to complete all study requirements
* Written informed consent obtained, including consent for tissue to be examined and stored by the central dermatopathologist
* Written consent to allow photographs of the target SCCIS lesion to be used as part of the study data
* For females of childbearing potential, a negative pregnancy test at screening and using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy)

Exclusion Criteria:

* Pregnant or lactating
* Presence of known or suspected systemic cancer
* Histological evidence of nBCC, sBCC, or any other tumor in the biopsy specimen
* Histological evidence of severe squamous metaplasia, infiltrative, desomoplastic or micronodular growth patterns in the biopsy specimen
* History of recurrence of the target SCCIS lesion
* Evidence of dermatological disease or confounding skin condition in the treatment area, e.g., BCC, actinic keratosis, rosacea, psoriasis, atopic dermatitis, eczema, xeroderma pigmentosa
* Concurrent disease or treatment that suppresses the immune system
* Chronic medical condition that in the judgment of the investigator(s) would interfere with the performance of the study or would place the patient at undue risk
* Known sensitivity to any of the ingredients in the study medication
* Use of a tanning parlor or other excessive or prolonged exposure to ultraviolet light or direct sunlight during the course of the study
* Treatment with systemic chemotherapeutic agents within the 6 months prior to the screening visit
* Use of systemic retinoids within the 6 months prior to the screening period
* Treatment with systemic immunomodulators or immunosuppressants within the 6 months prior to the screening period
* Use of topical immunomodulators within 2 cm of the target SCCIS lesion within the 4 weeks prior to the screening period
* Treatment with the following topical agents within the 4 weeks prior to the screening visit: levulanic acid, 5-fluorouracil, corticosteroids, retinoids, diclofenac, hyaluronic acid, imiquimod
* Undergone a facial resurfacing procedure, i.e., chemical peel, laser resurfacing, dermabrasion, within the 6 months prior to the screening visit, if the target SCCIS lesion is on the face
* Treatment with liquid nitrogen, surgical excision or curettage within 2 cm of the target SCCIS lesion during the 4 weeks prior to the screening visit
* Elective surgery within 4 weeks prior to the screening visit, during the study, or 4 weeks after the treatment period
* Evidence of current chronic alcohol or drug abuse
* Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of the screening visit
* In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions of the protocol and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the proportion of subjects with a complete response for the Intent-to-Treat (ITT) population. | 8 weeks

SECONDARY OUTCOMES:
The secondary efficacy endpoint is the proportion of subjects with a partial response in the ITT population. | 8 weeks